CLINICAL TRIAL: NCT03353051
Title: Iron and Infection: Neonatal Nutritional Immunity (NeoInnate Study)
Brief Title: Iron and Infection: Neonatal Nutritional Immunity
Acronym: NeoInnate
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Oxford (Other); Department of State for Health and Social Welfare, The Gambia (Other Government)
Responsible Party: Sponsor
Other Study IDs: SCC1525
Record Dates: First submitted 2017-07-20; First posted 2017-11-27 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Neonatal Infection; Nutritional Anemia
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be kept for follow up analysis if further iron and inflammation parameters require quantification.
  G6PD deficiency and sickle cell disease are confounders in the bacterial growth assay. G6PD deficiency genetic test will be performed on whole blood. Sickle cell will be assessed by PCR. Samples will be saved for additional possible DNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group A: other - observational study: neonates ≥2000-<2500g and born with a gestation age <37 weeks.
  Interventions: Other: Observational study
- Group B: other- observational study: Group B will contain neonates >2500g and born with a gestation age <37 weeks.
  Interventions: Other: Observational study
- Group C: other - observational study: Group C will contain neonates ≥2000-<2500g but with a gestation age >37 weeks.
  Interventions: Other: Observational study
- Group D1:other - observational study: Neonate >2500g and born with a gestation age >37 weeks. These neonates will donate blood at 6-24hrs and at 30-48hrs.
  Interventions: Other: Observational study
- Group D2: other - observational study: Neonate >2500g and born with a gestation age >37 weeks. These neonates will donate blood at 6-24hrs and at 42-60hrs
  Interventions: Other: Observational study
- Group D3: other - observational study: Neonate >2500g and born with a gestation age >37 weeks. These neonates will donate blood at 6-24hrs and at 144-192hrs.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
The motivation for this study was produced from our preliminary data, which showed that during the first 96 hours of life a full-term neonate will actively reduce the overall serum iron concentration of their blood and the transferrin saturation decreases rapidly from 45% in cord blood to ~20% by six hours post-delivery.

The Investigators hypothesise that this active sequestration of iron, which results in hypoferremia, is done in an effort to limit susceptibility to infection, a process referred to as nutritional immunity.

Currently, little is known about iron regulation and iron homeostasis during the first week of life and even less is known about the comparisons of nutritional immunity between full term, preterm and low birth weight neonates. Additionally, limited research has been conducted on the impact of these processes on bacterial pathogens.

In an effort to study the neonatal nutritional immunity and its role in neonatal susceptibility to infection, The investigator will conduct an observational study in full-term, preterm and low birth weight vaginally-delivered neonates born at Serrekunda General Hospital, The Gambia.

The investigators will fully characterise and quantify nutritional immunity during the early neonatal period and the investogators will assess how this impacts bacterial growth. Study sensitisation will occur at the antenatal clinic, during the mother's second trimester of pregnancy. Mothers will be consented and enrolled at delivery. Blood samples will be collected once from the umbilical cord and at serial time points from the neonates over the first week of life.

DETAILED DESCRIPTION:
The epicentres of neonatal death worldwide are West and Central Africa, with an estimated 35 deaths per 1000 births. Neonatal infection is the third largest cause of death in children under five worldwide and is an ongoing major global public health challenge (WHO Millennium Development Goal 4). Intrauterine and neonatal infections have a high risk of causing substantial long-term neurological morbidity, affecting not just the individual but the local community and national productivity. Current research on neonatal sepsis in low-resource settings is focused on the use of mass perinatal antibiotic therapy for both mothers and babies. However, antibiotic resistance in the developing world is dramatically increasing and ablation of the neonatal microbiome has been linked with long-term health consequences. Novel therapeutic solutions are urgently required.

Nutritional immunity is the process by which the host innate immune system limits nutrient availability to invading organisms. Iron is an essential micronutrient for both microbial pathogens and their mammalian hosts. Changes in iron availability and distribution have significant effects on pathogen virulence and on the immune response to infection. Commonly found in blood, iron and its moieties (heme) are sequestered mainly in chaperone molecules (transferrin, lactoferrin, haptoglobin, hemopexin). The long-term goal of our research is to develop an anti-virulence therapeutic strategy that will augment nutritional immunity in the at-risk newborn, in order to improve neonatal survival, while avoiding the use of traditional empirical antibiotics.

During the dynamic neonatal period there are significant changes in circulation, oxygenation and iron homeostasis, the foetus maintains a high haematocrit to facilitate perfusion in utero. Within the first week of life, the neonate's haematocrit decreases as the RBCs containing foetal haemoglobin are broken down. Our preliminary data shows that during the first 24 hours of life full-term neonates will actively reduce the overall serum iron concentration and transferrin saturation decreases rapidly from 45% in cord blood to ~20% by six hours post-delivery.

Currently, little is known about nutritional immunity in the neonates or about its impact on bacterial pathogens. In the aims below, the investigators will investigate the hypothesis that nutritional immunity may be an evolutionary mechanism designed to protect neonates from infection during the first critical days of life, by limiting the pathogenicity and virulence of these organisms by reducing the availability of iron. The investigators hypothesize that this protective mechanism may not be activated in preterm and low birth weight neonates, putting these babies at an enhanced risk of neonatal infection.

Host chaperoned or unchaperoned iron, hemoglobin and heme in the blood can provide a growth-limiting nutrient to bacterial pathogens depending on the specific bacterial species and their iron-uptake mechanisms. Bacterial co-evolution with the host has resulted in two main strategies to combat host nutritional immunity: (1) chelation of iron away from chaperone proteins with siderophores, and (2) direct uptake of hemoglobin and heme moieties. Previous research and preliminary experiments conducted by our group, using ex-vivo growth assays in adult serum, has shown that growth of a panel of neonatal pathogenic bacteria each decreases in response to decreasing transferrin saturation and increases in response to increasing hemoglobin concentration. In addition, the investigators have shown that the in vitro growth of standard laboratory strains of four important causes of early neonatal sepsis in the developing world (Staphylococcus aureus, Klebsiella pneumoniae, Escherichia coli, and Streptococcus agalactiae) is decreased in hypoferremic serum collected from full term neonates between 6-24 hours after birth compared to serum from the umbilical cord at birth.

In an effort to study neonatal nutritional immunity and its role in neonatal susceptibility to infection, the investigators will conduct an observational study in full-term (FT), preterm (PTB) and low birth weight (LBW) vaginally-delivered neonates born at Serrekunda Hospital in The Gambia. The investigators will fully characterize and quantify nutritional immunity during the early neonatal period (Research Question 1, Research Question 2 and Research Question 3) and the investigators will assess how it impacts bacterial growth using in vitro assays (Research Question 4). Mothers will be consented and enrolled at delivery. Blood samples will be collected once from the umbilical cord and at serial time points from the neonates (see sampling schema).

ELIGIBILITY:
Inclusion Criteria:

Low Birth Weight (LBW) neonates:

* Medical stable neonates
* Neonatal weight ≥2000g and <2500g
* Born at Serrekunda Hospital
* Gestational age will be >37 weeks.
* Born to mothers at least 18 years of age

Preterm neonates with Low Birth Weight (PTB+LBW):

* Medical stable neonates
* Born at Serrekunda Hospital
* Neonates weighing <2500g and <37 weeks of gestational age.
* Born to mothers at least 18 years of age

Preterm (PTB) neonates:

* Medical stable neonates
* >32 and <37 weeks' gestational age
* Born at Serrekunda Hospital
* PTB neonates will weigh more than 2500g
* Born to mothers at least 18 years of age

Full Term (FT) neonates:

* Healthy neonates
* Born at Serrekunda Hospital
* FT neonates will weigh ≥2500g
* Gestational age ≥37 weeks
* Born to mothers at least 18 years of age

Exclusion Criteria:

* Major congenital malformations
* Severe birth asphyxia
* Children from multiple births
* Medication (i.e. prophylactic antibiotics) given to neonate before first neonatal venous blood draw
* Neonates born via Breech, Vacuum or C section
* Neonates with infection/illness (information gained from venous bleed) will no longer be required to give future samples if originally required

Ages: 5 Minutes to 28 Days | Sex: All
Age Groups: Child
Study Population: All neonates will be born at Serrekunda Hospital, The Gambia. New Ballard score is only measure used to evaluate gestational age
  Preterm neonates with Low Birth Weight (PTB with LBW) (Group A): Neonates will not be recruited directly into this group. These medical stable neonates will weigh <2500g and also be <37 weeks of gestational age.
  Preterm (PTB) neonates (Group B): Medical stable neonates between >32 and <37 weeks' gestational age. PTB neonates will weigh >2500g.
  Low Birth Weight (LBW) neonates (Group C): Medical stable neonates with weight equal to or >2000g and <2500g. LBW neonates will have a gestational age of >32 weeks.
  Full Term (FT) neonates (Group D1-D3): All healthy FT neonates will weigh ≥2500g with gestational age ≥37 weeks.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
serum iron | at 7 days after birth
  will be measured using a COBAS INTEGRA 400 plus clinical chemistry analyzer

SECONDARY OUTCOMES:
TSAT (%) and heme iron (mg/dL) | at 6 hours after birth
  During the neonatal transition period in PTB and LBW neonates and FT babies in cord blood and at 6 hours after birth. TSAT and heme iron will be measured using a using a COBAS INTEGRA 400 plus clinical chemistry analyzer .
Iron (ug/dL), TSAT (%) and heme iron (mg/dL) regulated regulation in FT neonates | 7 days after birth
  During the first 7 days of life. Iron, TSAT and heme iron will be measured using a using a COBAS INTEGRA 400 plus clinical chemistry analyzer
microorganisms that are common causes of neonatal sepsis | At 0, 6 and 24 hours after birth
  Does sera from PTB and LBW neonates after birth support more ex-vivo growth of microorganisms that are common causes of neonatal sepsis in Africa and The Gambia (Staphylococcus aureus, Klebsiella pneumoniae, Escherichia coli, Group B Streptococcus, Streptococcus pneumoniae and Salmonella Tyhpimurium) than sera from FT neonates

CONTACTS AND LOCATIONS:
Overall Officials: Carla Cerami, MD, PhD, Principal Investigator — Medical Council Unit the Gambia
Locations (1):
- Serrekunda General Hospital, Kanifing, Near Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cross JH, Jarjou O, Mohammed NI, Gomez SR, Touray BJB, Kessler NJ, Prentice AM, Cerami C. Iron homeostasis in full-term, normal birthweight Gambian neonates over the first week of life. Sci Rep. 2023 Jun 26;13(1):10349. doi: 10.1038/s41598-023-34592-z. PMID 37365154
- [Derived] Cross JH, Jarjou O, Mohammed NI, Rayment Gomez S, Touray BJB, Prentice AM, Cerami C. Early postnatal hypoferremia in low birthweight and preterm babies: A prospective cohort study in hospital-delivered Gambian neonates. EBioMedicine. 2020 Feb;52:102613. doi: 10.1016/j.ebiom.2019.102613. Epub 2020 Jan 22. PMID 31981986
- [Derived] Cross JH, Jarjou O, Mohammed NI, Prentice AM, Cerami C. Neonatal iron distribution and infection susceptibility in full term, preterm and low birthweight babies in urban Gambia: study protocol for an observational study. Gates Open Res. 2019 Oct 15;3:1469. doi: 10.12688/gatesopenres.12963.2. eCollection 2019. PMID 31588425